CLINICAL TRIAL: NCT05457946
Title: A Prospective, Multi-national, Multi-center, Open-label, Randomized, Active-controlled, Parallel-group, Operationally Seamless Phase 2/3 Clinical Study to Evaluate the Immunogenicity and Safety of LBVD, a Fully Liquid Hexavalent Diphtheria-Tetanus-Whole Cell Pertussis-Hepatitis B-poliomyelitis (Inactivated)-Haemophilus Influenzae Type b Conjugate (DTwP-HepB-IPV-Hib) Vaccine, Given to Healthy Infants at 6-, 10-, and 14-week of Age as Primary Series
Brief Title: Study to Evaluate the Immunogenicity and Safety of LBVD(Hexavalent Vaccine), Given to Healthy Infants at Primary Series
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LG-VDCL003
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Diphtheria; Tetanus; Pertussis; Hepatitis B; Poliomyelitis; Haemophilus Influenzae Type B Infection
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Hepatitis B; Poliomyelitis; Haemophilus Infections | interventions — Vaccines, Combined; Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Test group 1 (Experimental): Low dose of candidate hexavalent vaccine (DTwPHepB-Sabin IPV-Hib) for Stage 1/ selected dose of hexavalent vaccine Lot A for Stage 2
  Interventions: Biological: LBVD (Hexavalent vaccine)
- Test group 2 (Experimental): Middle dose of candidate hexavalent vaccine (DTwPHepB-Sabin IPV-Hib) for Stage 1/ selected dose of hexavalent vaccine Lot B for Stage 2
  Interventions: Biological: LBVD (Hexavalent vaccine)
- Test group 3 (Experimental): High dose of candidate hexavalent vaccine (DTwPHepB-Sabin IPV-Hib)for Stage 1/ selected dose of hexavalent vaccine Lot C for Stage 2
  Interventions: Biological: LBVD (Hexavalent vaccine)
- Control group (Active Comparator): Co-administration of Pentavalent vaccine and Inactivated Polio vaccine for both stages
  Interventions: Biological: Pentavalent vaccine and Inactivated Polio vaccine (Sabin strains)

INTERVENTIONS:
Biological: LBVD (Hexavalent vaccine) — Injection within the muscle into the front area of the thigh
  Arms: Test group 1; Test group 2; Test group 3
Biological: Pentavalent vaccine and Inactivated Polio vaccine (Sabin strains) — Injection within the muscle into the front area of the thigh
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate immunogenicity and safety of different doses of candidate hexavalent vaccine in comparison to co-administration of Pentavalent vaccine and Poliomyelitis Vaccine (Inactivated) in separate injections at four weeks after completion of three-dose primary series at 6-10-14 weeks of age when administered to healthy infants and thereby to select the optimal dose of candidate vaccine(Stage 1) and to demonstrate lot-to-lot consistency of three lots of LBVD (Stage 2)

DETAILED DESCRIPTION:
Stage 1 (Dose-level Finding;Phase 2)

1. To compare the immunogenicity and safety of three LBVD vaccine candidates, varying at different dose levels, to the Control vaccines at 4 weeks after a three-dose primary series of vaccination and thereby, select an optimal vaccine dose level for Stage 2

Stage 2 (Evaluation of Safety, Immunogenicity, and Lot-to-lot Consistency;Phase 3)

1. To demonstrate the non-inferiority and lot-to-lot consistency in the immunogenicity of three separate lots of LBVD to the Control vaccines at 4 weeks after a three-dose primary series of vaccination given at 6-, 10- and 14-week of age
2. To demonstrate the safety and immunogenicity of LBVD at 4 weeks after a three-dose primary series of vaccination given at 6-, 10- and 14-week of age

ELIGIBILITY:
Inclusion Criteria:

* Infants in stable health
* Male or female 6 to 8 weeks of age
* Signed informed consent by the infant's parent(s) or legally acceptable representative(s)

Exclusion Criteria:

* Known or suspected Hib, HepB, diphtheria, tetanus, pertussis, or poliomyelitis
* Fever ≥ 38.0℃/100.4℉ within 3 days prior to study registration
* Known or suspected immunodeficiency
* Previous use of blood or blood-derived products
* Previous use of any diphtheria, tetanus, pertussis-based combination vaccine(s), Hib conjugate, poliovirus, or combination
* Household contact or intimate exposure with a confirmed case of Hib, HepB, diphtheria, pertussis, tetanus or poliomyelitis within 30 days prior to study registration
* Any history of allergy (hypersensitivity) to any of the vaccine components
* Participation in another interventional clinical trial simultaneously

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1438 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Seroprotection/seroconservison/ vaccine-response rate | 4 weeks after three-dose primary series
  Proportion of subjects achieving seroprotection/seroconversion/vaccine-response to each antigenic components

SECONDARY OUTCOMES:
Geometric mean concentration (GMC) or Geometric mean titer (GMT) | 4 weeks after three-dose primary series
  GMC or GMT and their ratio of all types of antibodies
Immediate reactions after vaccination | 30 minutes after each vaccination
  Immediate reactions after vaccination including all the signs and symptoms that occur within 30 minutes after the vaccination will be monitored at site. It is collected as an adverse event, but is classified as an immediate reaction only if the AE occurs within 30 minutes after vaccination.
Solicited adverse event | 7 days after each vaccination
  Expected local or systemic side effects after vaccination
Unsolicited adverse event | 28 days after each vaccinations
  All unwanted or bad events after vaccination other than solicited adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Edison Alberto, MD, Principal Investigator — Health Index Multispecialty Clinic; Josefina Carlos, MD, Principal Investigator — UERM Memorial Medical Center